CLINICAL TRIAL: NCT01028482
Title: Treatment of Postpartum Depression With Psychotherapy and Add-on Sertraline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Miki Bloch MD, Tel aviv Sourasky medical center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-09-MB-301-CTIL
Record Dates: First submitted 2009-06-03; First posted 2009-12-09 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Postpartum Depression
Keywords: severity of depression measured by MADRS and CGI
MeSH Terms: conditions — Depression, Postpartum | interventions — Sertraline; Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sertraline, psychotherapy (Experimental): both study groups will receive concomitant psychotherapy treatment. There will be 2 main comparison groups: 1) an sertraline treated group and 2) a drug placebo - controlled group. While this design lacks a blinded "drug-only" condition, we will have an "open" drug-only arm that will be of considerable value. Furthermore, while a true placebo group is also lacking, and a certain response to psychotherapy is expected, we believe that the drug condition will show a definite superiority to the psychotherapy + placebo condition. The rational for including psychotherapy in the treatment protocol is the fact that this is a well-established treatment for PPD, and for ethical considerations it is unreasonable not to administer any active treatment to women suffering from PPD. It is our conviction that this is the only design, albeit its limitations, which will allow a comparison between medication-treated vs. placebo-treated PPD patients.
  Interventions: Drug: Sertraline; Other: psychotherapy
- placebo, psychotherapy (Placebo Comparator): both study groups will receive concomitant psychotherapy treatment. There will be 2 main comparison groups: 1) an sertraline treated group and 2) a drug placebo - controlled group. While this design lacks a blinded "drug-only" condition, we will have an "open" drug-only arm that will be of considerable value. Furthermore, while a true placebo group is also lacking, and a certain response to psychotherapy is expected, we believe that the drug condition will show a definite superiority to the psychotherapy + placebo condition. The rational for including psychotherapy in the treatment protocol is the fact that this is a well-established treatment for PPD, and for ethical considerations it is unreasonable not to administer any active treatment to women suffering from PPD. It is our conviction that this is the only design, albeit its limitations, which will allow a comparison between medication-treated vs. placebo-treated PPD patients.
  Interventions: Drug: placebo; Other: psychotherapy

INTERVENTIONS:
Drug: Sertraline — group A- sertraline 50-100 mg/day and weekly psychotherapy for 3 months
  group B- weekly psychotherapy- for 3 months
  group C- sertraline 50-100 mg/day-for 3 months
  Arms: sertraline, psychotherapy
Drug: placebo — placebo
  Arms: placebo, psychotherapy
Other: psychotherapy — psychotherapy

SUMMARY:
Introduction:

Postpartum depression (PPD) occurs in large numbers of women (between 10 - 20%) and substantially affects both their own well-being and their offspring's mental and emotional development. Whereas PPD is a form of major depression, its etiology is probably related to a combination of biological (hereditary, hormonal etc.), and psychological factors. In practice, most women suffering from PPD do not seek treatment, or are treated with psychotherapy alone due to concerns regarding pharmacotherapy. This is despite the obvious importance of reaching a rapid remission in these women. In fact, data regarding the treatment of PPD with antidepressants is surprisingly sparse and is limited to only one blinded and placebo-controlled study (with fluoxetine) and a number of studies without a placebo arm . The reason for the paucity of double-blinded placebo-controlled studies is probably due to 3 main limiting factors: Firstly, the reluctance of women to "admit" to and seek professional help due to depression, Secondly, the difficulty to administer antidepressant medication to lactating women, and, Thirdly, the ethical difficulties in designing a study with a real placebo group.

In contrast to the very limited number of drug studies in this population, there are a number of studies that have shown the efficacy of psychotherapy in the treatment of PPD. Positive studies have been published using different types of psychotherapy, including cognitive, dynamic and interpersonal psychotherapy.

The investigators propose to study the efficacy of psychotherapeutic treatment in women suffering from PPD with add-on sertraline in a randomized double-blind, placebo-controlled design. To overcome the difficulties described above in studying antidepressants in the postpartum period, the investigators propose to include active brief dynamic psychotherapy for all women. Furthermore, the investigators will selectively allow inclusion of women who only suffer from either mild or moderate major PPD (not severe / suicidal) .

Hypothesis:

The investigators hypothesize that women with PPD randomized to the arm receiving psychotherapy + active sertraline will show a greater response rate than the psychotherapy + placebo group. Furthermore, the investigators hypothesize that the difference in response between the 2 groups will demonstrate a significant early response in the active sertraline group.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18- 45 y.o.
2. SCID-DSM-IV diagnosis of major depression, mild to moderate severity
3. Understanding of Hebrew
4. Willing to sign the informed consent
5. Lactating women will be included after a thorough explanation of current knowledge of sertraline and lactation.

Exclusion Criteria:

1. Severe major depression (MADRS > 30)
2. Suicidal ideation (MADRS item 10 score of > 5)
3. Psychotic symptoms or aggressive thoughts toward the baby.
4. Current treatment with antidepressant medication
5. Physical illness explaining depressive symptoms (e.g. hypothyroidism, neurological disease, severe anemia, renal failure etc.)
6. Alcoholism or drug abuse and dependence
7. Bipolar Disorder
8. Past severe side effects to SSRIs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2008-03; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
depression | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Bloch M, Meiboom H, Lorberblatt M, Bluvstein I, Aharonov I, Schreiber S. The effect of sertraline add-on to brief dynamic psychotherapy for the treatment of postpartum depression: a randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2012 Feb;73(2):235-41. doi: 10.4088/JCP.11m07117. PMID 22401479